CLINICAL TRIAL: NCT01374035
Title: Interface Between Primary Care and Specialist Mental Health Care - the Referral Letters
Brief Title: The Western Norway Mental Health Interface Study on Referral Letters
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Were not able to conduct the intervention.
Sponsor: Helse Fonna (Other)
Collaborators: University of Bergen (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Miriam Hartveit, PhD-student, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NSD-24340
Record Dates: First submitted 2011-04-28; First posted 2011-06-15 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Mental Disorders
Keywords: Health Service; Coordination; Referral letters; Mental Health; Adults
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participating GPs (Experimental): GPs working at randomly selected GP centers/offices within the region that are invited to participate and signs a written informed consent to participate. (N=30-40)
  Interventions: Other: Quality improvement intervention
- Control group (No Intervention): GPs working at randomly selected GP centers/office within the region that are not invited to participate, will form the control group. (N=30-40)

INTERVENTIONS:
Other: Quality improvement intervention — A complex intervention will be implemented within the group of GPs in the intervention group. It includes participation in defining criteria for good referral letters, information about the correlation between information in the referral letters and outcome, introduction to the guideline, and consecutive feedback on own preformance regarding content of referral letter and outcome for the patient.
  Arms: Participating GPs

SUMMARY:
The main object to this trial is to study the function of referral letters as a mean to coordinate the care process for adult people when referred from Primary Care to Specialised Mental Health Care. The study will explore if and to what degree the quality of these referral letters can be improved, and the potential improvement's impact on defined patient-, professional and organisational related outcomes. According to Medical Research Council guidelines for evaluating complex interventions, a stepwise design with the use of both qualitative and quantitative methods will be used to conduct a controlled intervention study.

DETAILED DESCRIPTION:
The study is based on a stepwise progression including four steps. Within step one group interview with four mixed groups of health professionals (both Primary and Specialised Care), patient representatives and managers will be conducted. The groups will give input on firstly, what information they think is important to include in the referral letters, and secondly, what impact they think improved referral letters can have for the organisation and care within Specialised Mental Health Care. Within step two a validated check-list to assess the quality of referral letters will be developed. Within step three outcome measures will be developed and tested. Both step two and three will make use of the results from step one in addition to existing literature and testing. Step four is the intervention study where measures from the former steps will be used.

ELIGIBILITY:
Inclusion Criteria:

* Referral letters send from a GP to Public Specialised Mental Health Care
* Referrals for elective assessment or treatment

Exclusion Criteria:

* Referral letters send from other health personnel
* Referrals for acute care (within 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Length of stay | Day of discharge assessed up to six months
  From date of admission or onset of out-patient treatment until date of discharge (documented in Electronic Patient Record as end of treatment periode), assessed up to six months from admission.

SECONDARY OUTCOMES:
Response time for referral letters in Specialised Mental Health Care | Referral letters will be followed for the duration of the assessment and prioritation process until response letter is sent, an expected avarage of 10 days.
  Unit of measure: Number of days from receiving a referral letter to the response letter is sent to the patient and the General Practitioner. The response time for all letters recieved in a six month periode before the intervention to improve the quality of referral letters will be compared with the response time after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aslak B Aslaksen, MD, PhD, Study Chair — Faculty of Medicine and Dentistery, University of Bergen, Norway; Kjell Haug, MD, PhD, Principal Investigator — Faculty of Medicine and Dentistery, University of Bergen, Norway; Kris Vanhaecht, RN, PhD, Principal Investigator — KU Leuven
Locations (1):
- Helse Fonna Local Health Authorities, Haugesund, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartveit M, Biringer E, Vanhaeht K, Haug K, Aslaksen A. The Western Norway mental health interface study: a controlled intervention trial on referral letters between primary care and specialist mental health care. BMC Psychiatry. 2011 Nov 14;11:177. doi: 10.1186/1471-244X-11-177. PMID 22081994
- [Background] Hartveit M, Aslaksen A, Vanhaecht K, Thorsen O, Hove O, Haug K et al. Development and testing of an instrument in Western Norway to measure the quality of referral information from primary care to specialised mental health care. International Journal of Care Coordination18:2-3, 2015
- [Background] Hartveit M, Vanhaecht K, Thorsen O, Biringer E, Haug K, Aslaksen A. Quality indicators for the referral process from primary to specialised mental health care: an explorative study in accordance with the RAND appropriateness method. BMC Health Serv Res. 2017 Jan 3;17(1):4. doi: 10.1186/s12913-016-1941-1. PMID 28049470
- [Result] Hartveit M, Thorsen O, Biringer E, Vanhaecht K, Carlsen B, Aslaksen A. Recommended content of referral letters from general practitioners to specialised mental health care: a qualitative multi-perspective study. BMC Health Serv Res. 2013 Aug 19;13:329. doi: 10.1186/1472-6963-13-329. PMID 23958371
- [Derived] Nymoen M, Biringer E, Hetlevik O, Thorsen O, Assmus J, Hartveit M. The impact of referral letter quality on timely access to specialised mental health care: a quantitative study of the reliability of patient triage. BMC Health Serv Res. 2022 Jun 2;22(1):735. doi: 10.1186/s12913-022-08139-3. PMID 35655302